CLINICAL TRIAL: NCT03767270
Title: A Phase 1/2 Single Ascending Dose Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenously Administered MRT5201 in Subjects With Ornithine Transcarbamylase Deficiency
Brief Title: Safety, Tolerability and PK/PD Evaluation of Intravenous Administration of MRT5201 in Patients With OTC Deficiency
Acronym: STEP-OTC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Program was discontinued.
Sponsor: Translate Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRT5201-101; 2018-004095-35 (EudraCT Number)
Record Dates: First submitted 2018-11-28; First posted 2018-12-06 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Ornithine Transcarbamylase Deficiency
Keywords: OTC; Urea Cycle Disorder; UCD
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease; Urea Cycle Disorders, Inborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MRT5201 (Experimental): Single Ascending Low, Mid, and High doses of MRT5201
  Interventions: Biological: MRT5201
- Placebo (Placebo Comparator): Placebo comparator using 5% dextrose in water at the same administration rate as study drug.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MRT5201 — Codon-optimized human ornithine transcarbamylase messenger ribonucleic acid with lipid-based nanoparticles
  Arms: MRT5201
Other: Placebo — 5% dextrose in water
  Arms: Placebo

SUMMARY:
This Phase 1/2, first-in-human study will evaluate the safety and tolerability of single escalating doses of MRT5201 administered intravenously to subjects with OTC Deficiency (OTCD). This study will also evaluate the effect of a single dose of MRT5201 on metabolic markers of OTCD and ureagenesis; and determine an acceptable dosing interval of MRT5201.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of OTCD.
* Documented history of ≥1 symptomatic hyperammonemia event with ammonia ≥100 µmol/L
* Subject's OTCD is stable as evidenced by meeting the following criteria:

  * Ammonia level <175 µmol/L during the Screening Period and at Baseline (Day -1)
  * No clinical symptoms of hyperammonemia during the Screening Period and at Baseline (Day -1)
* If using nitrogen scavenger therapy, must be on a stable regimen for ≥28 days prior to signing informed consent
* Subject has maintained a stable protein restricted diet (which may or may not include medical foods) and/or amino acid supplementation with no changes in calorie or protein goals and no changes in medical food and/or amino acid supplementation for ≥ 28 days prior to signing informed consent.

Exclusion Criteria:

* Any laboratory abnormality that may put the subject at increased risk by participating in this study.
* Have any significant concurrent or past medical condition that would represent an unacceptable risk to the subject or might jeopardize the collection of high-quality data from the study. These include but are not limited to:

  * History of liver transplant, including hepatocyte therapy/transplant
  * History of liver disease
  * Positive viral serology test results for HIV type 1 or 2 antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody
  * Type I or Type II diabetes that is poorly controlled, in the opinion of the Investigator
  * Poorly controlled hypertension (defined as systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 90 mm Hg)
  * Use of anticoagulants or platelet inhibitors, including but not limited to heparin and non-steroidal anti-inflammatory drugs (NSAIDS). Acetaminophen is permitted
* Participation in previous clinical studies evaluating investigational OTCD therapies directed at expressing functional OTC protein (eg, OTC gene therapy studies, other mRNA replacement therapy) that has led to the presence of anti-OTC antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment-emergent adverse events by treatment group | Week 24
  The incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) for each dosing cohort by treatment group, assessed by severity and relationship to study product.

SECONDARY OUTCOMES:
Pharmacokinetics parameters of MRT5201 | 1 month after single dose
  Pharmacokinetics of MRT5201 as measured by levels of mRNA
Effect of a single dose of MRT5201 on ureagenesis | Up to 1 month after single dose
  Change from Baseline in 4-hour ureagenesis AUC at weeks 2, 3, 4, and 5 after a single dose of MRT5201
Effect of single dose of MRT5201 on metabolic markers of OTCD | 6 months after single dose
  Change from Baseline in 8-hour ammonia AUC

IPD SHARING:
Plan to Share IPD: Undecided